CLINICAL TRIAL: NCT00003170
Title: Phase III Double-Blind Study of Glutamine Versus Placebo in the Prevention of Acute Diarrhea in Patients Receiving Pelvic Radiation Therapy
Brief Title: Glutamine in Preventing Acute Diarrhea in Patients With Pelvic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-969256; CDR0000065974 (Registry Identifier: PDQ (Physician Data Query)); NCI-P97-0127
Record Dates: First submitted 1999-11-01; First posted 2004-09-06 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glutamine (Experimental): Beginning the first or second day of radiotherapy, patients receive oral glutamine twice daily, including the days that they do not receive radiotherapy. Patients continue on treatment throughout radiotherapy and continue 2 weeks postradiotherapy or until grade 3 diarrhea occurs. Patients are followed weekly for 4 weeks, then at 12 months, and then at 24 months after radiotherapy.
  Interventions: Dietary Supplement: glutamine
- placebo (Placebo Comparator): Beginning the first or second day of radiotherapy, patients receive placebo twice daily, including the days that they do not receive radiotherapy. Patients continue on treatment throughout radiotherapy and continue 2 weeks postradiotherapy or until grade 3 diarrhea occurs. Patients are followed weekly for 4 weeks, then at 12 months, and then at 24 months after radiotherapy.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: glutamine
  Arms: glutamine
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Glutamine may be an effective treatment for acute diarrhea caused by radiation therapy. It is not known if glutamine is an effective treatment for acute diarrhea caused by radiation therapy.

PURPOSE: Randomized double-blinded phase III trial to determine the effectiveness of glutamine in preventing acute diarrhea in patients who have pelvic cancer and who are receiving radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether glutamine is effective in reducing the acute treatment related diarrhea in patients receiving pelvic external beam radiation therapy as adjuvant or primary treatment of malignancy. II. Determine whether glutamine can reduce chronic treatment related enteropathy following completion of therapy. III. Determine whether glutamine causes any toxicity in this situation. IV. Provide initial reliability and validity data for a patient bowel function questionnaire.

OUTLINE: This is a randomized, double-blind, placebo controlled study. Patients are stratified by history of anterior resection of the rectum (yes vs no); total planned cumulative dose, including boost fields of external beam radiotherapy (4500-5350 cGy vs 5350-6000 cGy vs greater than 6000 cGy); use of fluorouracil (none vs bolus vs continuous infusion); and primary site (rectal cancer vs prostate cancer vs gynecological cancer vs other). Beginning the first or second day of radiotherapy, patients receive either oral glutamine or a placebo twice daily, including the days that they do not receive radiotherapy. Patients continue on treatment throughout radiotherapy and continue 2 weeks postradiotherapy or until grade 3 diarrhea occurs. Patients are followed weekly for 4 weeks, then at 12 months, and then at 24 months after radiotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed pelvic cancer Planned therapy is to undergo continuous definitive or adjuvant external beam pelvic radiation therapy with or without fluorouracil (5-FU) plus or minus levamisole No split course radiation therapy Planned course of radiation therapy must also meet the following criteria: - Entire pelvis must be encompassed by the planned radiotherapy fields - Total planned dose to the central axis midplane or isocenter for the whole pelvic field must be between 4500-5350 cGy - Treatment must be given 4-5 times per week on a one-treatment-per-day basis No stool incontinence or stool frequency of 7 or more per day prior to initiation of radiation therapy Must be entered on study before the second radiation therapy fraction No current or prior metastases beyond pelvic regional lymph nodes Must have functioning rectum No planned perineal irradiation No anal cancer No active intraluminal gastrointestinal (GI) tumors Patients with completely resectioned GI tumors who also receive adjuvant treatment are eligible

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine less than 2 times upper limit of normal Other: No known allergy to glutamine No history of inflammatory bowel disease No other medical condition that may interfere with treatment Not pregnant or nursing Adequate contraception is required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent leucovorin or other chemotherapy agents, except 5-FU with or without levamisole Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior pelvic radiotherapy No brachytherapy prior to completion of all external beam radiotherapy Surgery: No abdominal-perineal resection, Hartmann procedure, or other surgical procedure that has left patient without a functioning rectum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 1998-02; Primary Completion 2003-05 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
reduction of acute treatment related to diarrhea | Up to 2 years post-radiation treatment
reduction of chronic treatment related to enteropathy | Up to 2 years post-radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F. Kozelsky, MD, Study Chair — Mayo Clinic
Locations (18):
- United States (17):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Kozelsky TF, Meyers GE, Sloan JA, Shanahan TG, Dick SJ, Moore RL, Engeler GP, Frank AR, McKone TK, Urias RE, Pilepich MV, Novotny PJ, Martenson JA; North Central Cancer Treatment Group. Phase III double-blind study of glutamine versus placebo for the prevention of acute diarrhea in patients receiving pelvic radiation therapy. J Clin Oncol. 2003 May 1;21(9):1669-74. doi: 10.1200/JCO.2003.05.060. PMID 12721240